CLINICAL TRIAL: NCT06211387
Title: ADDITIVE BENEFITS of KALTENBORN SUSTAINED STRETCH JOINT MOBILIZATION with RESISTANCE EXERCISE TRAINING in KNEE OSTEOARTHRITIS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/22
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance exercise + joint mobilization (Experimental)
  Interventions: Procedure: Resistance Exercise Training; Procedure: Joint Mobilization
- Resistance Exercise (Active Comparator)
  Interventions: Procedure: Resistance Exercise Training

INTERVENTIONS:
Procedure: Resistance Exercise Training — Resistance Exercise Training for knee
Procedure: Joint Mobilization — Tibiofemoral and Patellofemoral Joint Mobilization
  Arms: Resistance exercise + joint mobilization

SUMMARY:
to determine the supplementary effects of Kaltenborn sustained stretch mobilization when combined with resistance training in the management of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

Grade I-III knee OA Both male and female nee osteoarthritis for at least 3 months knee pain no more than 8/10

Exclusion Criteria:

Malignancy Any additional Inflammatory disorders Infection Knee trauma lower limb fracture Lumbar radiculopathy or myelopathy knee surgery Intra-articular steroid therapy in the last 2 months Total knee replacement (TKR). Total hip replacement (THR). Any neurological disorder Any cardio-pulmonary complications Rheumatoid arthritis Septic arthritis Recent history of trauma Osteoporosis or osteomyelitis Grade IV osteoarthritis

-

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-02 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
Knee Pain | 4 weeks
  Knee Pain will be quantified using Numeric Pain Rating Scale (NPRS). NPRS is a 11 point scale form 0-10. Lower Score on NPRS signifies less pain, whereas higher score on NPRS signifies more pain.
Physical Function | 4 weeks
  To determine the physical function related to knee osteoarthritis Western Ontario and McMaster Universities Arthritis Index (WOMAC) will be used with a total of 24 items and a higher score on WOMAC signifies poor outcome.
Isometric Muscle Strength | 4 weeks
  Modified Sphygmomanometer will be used to measure isometric muscle strength of the muscles of the knee joint. A higher score signifies greater strength.
Functional Mobility strength | 4 weeks
  5 repetition sit to stand test will be used to determine functional mobility strength. Less time to complete the task signifies better outcome.
Cadence | 4 weeks
  Observational gait analysis will be used to determine cadence. A higher score signifies better outcome.
Gait velocity | 4 weeks
  Observational gait analysis will be used to determine cadence. A higher score signifies better outcome.
Stride length | 4 weeks
  Observational gait analysis will be used to determine cadence. A higher score signifies better outcome.
Knee range of motion (ROM) | 4 weeks
  Gonimeter will be used to measure knee range of motion.. A higher score signifies better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anas Hameed, Principal Investigator — Foundation University Islamabad; Muhammad Osama, Study Chair — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan